CLINICAL TRIAL: NCT04135560
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, FIRST-IN-HUMAN, LOCAL TOLERABILITY AND DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE-DOSE, TOPICAL ADMINISTRATION OF PF-07038124 TO HEALTHY PARTICIPANTS
Brief Title: A Study To Determine The Safety, Tolerability, Skin Irritation Potential, And PK Following Topical Application Of PF-07038124 In Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3941001; FIH Study of PF-07038124 (Other: Alias Study Number)
Record Dates: First submitted 2019-10-07; First posted 2019-10-22 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Dermatitis Atopic
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A Cohort 1 (1% Body Surface Area) (Experimental): Each participant in this cohort will receive both PF-07038124 0.06% and vehicle applied to the skin (1% Body Surface Area)
  Interventions: Drug: PF-07038124 and Vehicle
- Part B Cohort 1 (10% Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Part B Cohort 2 (10% Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Part B Cohort 3 (10% Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Part B Cohort 4 (10% Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Part B Cohort 5 (20% Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Part B Cohort 6 (10% Body Surface Area) (Experimental): Optional cohort of Japanese participants
  Interventions: Drug: PF-07038124 or vehicle

INTERVENTIONS:
Drug: PF-07038124 and Vehicle — PF-07038124 0.06% and vehicle Ointment BID applied to 1% Body Surface Area (BSA)
  Arms: Part A Cohort 1 (1% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 0.01% or vehicle Ointment QD applied to 10% BSA
  Arms: Part B Cohort 1 (10% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 0.01% or vehicle Ointment BID applied to 10% BSA
  Arms: Part B Cohort 2 (10% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 0.03% or vehicle Ointment BID applied to 10% BSA
  Arms: Part B Cohort 3 (10% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 0.06% or vehicle ointment BID applied to 10% BSA
  Arms: Part B Cohort 4 (10% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 safe concentration or vehicle ointment BID applied to 20% BSA
  Arms: Part B Cohort 5 (20% Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 safe concentration or vehicle BID applied to 10% BSA
  Arms: Part B Cohort 6 (10% Body Surface Area)

SUMMARY:
The purpose of this study is to evaluate the skin irritation potential of PF-07038124 ointment and vehicle (placebo) in Part A following multiple-doses applied topically to healthy participants. In Part B, the safety, tolerability, pharmacokinetic (PK), and skin irritation potential of PF-07038124 will be evaluated. In Part A, the highest concentration of 0.06% PF-07038124 will be applied to normal skin with a small surface area of 20 cm2 (0.1% body surface area [BSA]), while Part B will evaluate application of PF-07038124 and vehicle (placebo) to a surface area of 2000 cm2 (10% BSA) and 4000 cm2 (20% BSA). These data will provide support for clinical development in participants with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female participants of non-childbearing potential and/or male participants who, at the time of screening, must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD):
2. Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Participants enrolling as Japanese in Part B must have 4 biologically Japanese grandparents who were born in Japan.
5. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Participants who have any visible skin damage or skin condition (eg sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations) in or around the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction.
2. Participants who have a history of or have active AD/eczema/urticaria.
3. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
4. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
5. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
6. Acute disease state (unstable medical condition such as nausea, vomiting, fever or diarrhea, etc) within 7 days of Day 1.
7. Have undergone significant trauma or major surgery within 4 weeks of screening.
8. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. (Refer to Section 6.5 for additional details).
9. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
10. A positive urine drug test.
11. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
12. Baseline 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
13. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.5 × upper limit of normal (ULN);
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
14. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
16. History of serious adverse reactions or hypersensitivity to any topical drug; or known allergy to any of the test product(s) or any components in the test product(s) or history of hypersensitivity; or allergic reactions to any of the study preparations as described in the PF-07038124 IB.
17. Not willing to refrain from shaving, the use of depilatories or other hair-removal activities, antiperspirants, lotions, skin creams, fragrances or perfumes, or body oils (eg, baby oil; coconut oil), use of hair products, hair gels, and hair oil in the treatment areas for 48 hours prior to admission to the CRU and for the duration of the stay in the CRU.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Treatment Emergent Treatment-Related Adverse Evenst (AEs) | through study completion, up to 38 days
  Incidence and severity of local and systemic treatment emergent AEs and withdrawals due to treatment emergent AEs
Part A: Number of Adverse Events by Severity | through study completion, up to 38 days
  Incidence and severity of local and systemic treatment emergent AEs and withdrawals due to treatment emergent AEs
Part B: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | through study completion, up to 41 days
  Assessment of AEs, safety laboratory tests, vital signs (including blood pressure, pulse rate and temperature), cardiac telemetry and 12-lead ECGs.
  Incidence and severity of local skin irritation.
Part B: Number of Adverse Events by Severity | through study completion, up to 41 days
  Assessment of AEs, safety laboratory tests, vital signs (including blood pressure, pulse rate and temperature), cardiac telemetry and 12-lead ECGs.
  Incidence and severity of local skin irritation.

SECONDARY OUTCOMES:
Part B: Maximum Observed Plasma Concentration (Cmax) | Days 1 and 10
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Days 1 and 10
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Days 1 and 10
Plasma Decay Half-Life (t1/2) | Days 1 and 10
Average Concentration at Steady State (Cav) | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3941001